CLINICAL TRIAL: NCT00781911
Title: A Phase 2, Multicenter, Two Tier Study of IMC-A12 in Combination With Depot Octreotide in Patients With Metastatic, Well or Moderately Differentiated Carcinoid or Islet Cell Carcinoma
Brief Title: A Study of Cixutumumab (IMC-A12) in Islet Cell Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13929; CP13-0710 (Other: ImClone Systems); I5A-IE-JAEE (Other: Eli Lilly and Company)
Record Dates: First submitted 2008-10-27; First posted 2008-10-29 (Estimated); Results first posted 2018-04-18 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Carcinoma; Neuroendocrine Tumors
Keywords: Islet Cell; CARCINOMA, ISLET CELL; Octreotide; depot octreotide acetate; Insulin-Like Growth Factor (IGF) 1; Metastatic, Carcinoid or Islet Cell; Neuroendocrine Tumors
MeSH Terms: conditions — Carcinoma; Neuroendocrine Tumors; Carcinoma, Islet Cell; Neoplasm Metastasis; Carcinoid Tumor | interventions — cixutumumab; Octreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Carcinoid tumor (Experimental): Participants with carcinoid tumor will receive cixutumumab 10 mg/kg over 1 hour every 2 weeks. Treatment will continue until there is evidence of disease progression, intolerable toxicity, or other withdrawal criteria are met. Participants must be receiving depot octreotide at the time of enrolling into the study. Participants on stable doses of depot octreotide will continue to receive the same dose and schedule of their last regimen.
  Interventions: Biological: Cixutumumab; Drug: depot octreotide
- Islet cell carcinoma (Experimental): Participants with islet cell carcinoma will receive cixutumumab 10 mg/kg over 1 hour every 2 weeks. Treatment will continue until there is evidence of disease progression, intolerable toxicity, or other withdrawal criteria are met. Participants must be receiving depot octreotide at the time of enrolling into the study. Participants on stable doses of depot octreotide will continue to receive the same dose and schedule of their last regimen.
  Interventions: Biological: Cixutumumab; Drug: depot octreotide

INTERVENTIONS:
Biological: Cixutumumab — Participants will receive cixutumumab IV 10 mg/kg over 1 hour every 2 weeks. Treatment will continue until there is evidence of disease progression, intolerable toxicity, or other withdrawal criteria are met.
  Other Names: IMC-A12; LY3012217
Drug: depot octreotide — Participants must be receiving depot octreotide at the time of enrolling into the study. Participants on stable doses of depot octreotide will continue to receive the same dose and schedule of their last regimen.
  Other Names: SMS 201-995

SUMMARY:
Determine the 6-month progression free survival (PFS) rate associated with cixutumumab in combination with depot octreotide acetate (octreotide) in participants with metastatic neuroendocrine tumors.

ELIGIBILITY:
Inclusion Criteria:

* The participant has well-differentiated or moderately-differentiated, histologically confirmed neuroendocrine carcinoma, including carcinoid of any location and islet cell tumors
* The participant has metastatic disease at the time of study entry
* The participant must have a tumor measurable according to Response Evaluation Criteria in Solid Tumors (RECIST) guidelines, measurable by elevated tumor markers (eg, 24-hour urine 5-HIAA, chromogranin A, adrenocorticotropin hormone (ACTH), gastrin, or other tumor specific biochemical markers), or both
* The participant is age ≥ 18 years
* The participant's tumor has Ki-67 expression ≤ 20%
* The participant is receiving depot octreotide therapy at the time of enrolling into the study
* The participant has received 0 - 2 systemic anticancer regimens in addition to depot octreotide, which may have included chemotherapy, interferon, antiangiogenic therapy, other targeted treatments, or a combination of such treatments
* The participant is no longer a candidate for surgery, embolization, or radiofrequency ablation therapy
* The participant has experienced radiographic, biochemical, and/or scintigraphic disease progression while on a regimen that includes octreotide
* The participant has completed prior chemotherapy and/or radiotherapy with curative intent at least 3 weeks prior to the administration of the first dose of study therapy. Participants that have received palliative radiation therapy to bony metastases prior to the first dose of study medication are eligible
* The participant has a life expectancy of > 3 months
* The participant has an Eastern Cooperative Oncology Group performance status (ECOG PS) of 0-2
* The participant has adequate hematologic function as defined by absolute neutrophil count ≥ 1500/microliters (μL), hemoglobin ≥ 9 gram/deciliter (g/dL), and platelet count ≥100,000/μL
* The participant has adequate hepatic function as defined by a total bilirubin ≤ 1.5 x the upper limit of normal (ULN), and aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 3 x the ULN (or ≤ 5 x the ULN in the presence of known liver metastases)
* The participant either has adequate coagulation function as defined by international normalized ratio (INR) ≤ 1.5 and partial thromboplastin time (PTT) no more than 5 seconds above the ULN, or is on a stable dose of anticoagulant
* The participant has adequate renal function as defined by serum creatinine ≤ 1.5 x the institutional ULN or creatinine clearance ≥ 60 milliliter/minute (mL/min) for participants with creatinine levels above the ULN
* The participant has fasting serum glucose < 160 milligram/deciliter (mg/dL) and hemoglobin A1c (HgbA1c)≤ 7. If baseline nonfasting glucose is < 160 mg/dL, fasting glucose measurement is not required
* Because the teratogenicity of cixutumumab is not known, women of childbearing potential (WOCBP) must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation
* The participant has the ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* The participant has uncontrolled brain or leptomeningeal metastases
* The participant has not recovered to Grade ≤ 1 from adverse events due to agents administered more than 4 weeks prior to study entry (except for alopecia)
* The participant is receiving any other investigational agent(s)
* The participant has received therapeutic radiolabeled somatostatin analogues
* The participant has received more than 2 prior regimens of systemic therapy in the metastatic setting
* The participant has a history of treatment with other agents targeting the IGF receptor
* The participant has a history of allergic reactions attributed to compounds of chemical or biologic composition similar to that of cixutumumab or to octreotide
* The participant has poorly controlled diabetes mellitus. Participants with a history of diabetes mellitus are allowed to participate, provided that their fasting glucose < 160 mg/dL or below the ULN and that they are on a stable dietary or therapeutic regimen for this condition
* The participant has an uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring parenteral antibiotics, symptomatic congestive heart failure, uncontrolled hypertension, clinically significant cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* The participant is pregnant or lactating
* The participant is known to be positive for infection with the human immunodeficiency virus
* The participant has a history of another primary cancer, with the exception of: a) curatively resected nonmelanomatous skin cancer; b) curatively treated cervical carcinoma in-situ; or c) other primary solid tumor curatively resected or treated with no known active disease present and no treatment administered for the last 3 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2009-02; Primary Completion 2011-07 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (9):
- United States (9):
  - ImClone Investigational Site, Los Angeles, California
  - ImClone Investigational Site, Aurora, Colorado
  - ImClone Investigational Site, Atlanta, Georgia
  - ImClone Investigational Site, Indianapolis, Indiana
  - ImClone Investigational Site, Kenner, Louisiana
  - ImClone Investigational Site, Columbus, Ohio
  - ImClone Investigational Site, Providence, Rhode Island
  - ImClone Investigational Site, Nashville, Tennessee
  - ImClone Investigational Site, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who completed the study include those who died and had progressive disease.
Groups:
- Carcinoid Tumor: Participants with carcinoid tumor received cixutumumab 10 mg/kg intravenously (IV) over 1 hour every 2 weeks. Treatment continued until there is evidence of disease progression, intolerable toxicity, or other withdrawal criteria are met.
  Participants must be receiving depot octreotide at the time of enrolling into the study. Participants on stable doses of depot octreotide continued to receive the same dose and schedule of their last regimen.
- Islet Cell Carcinoma: Participants with islet cell carcinoma received cixutumumab 10 mg/kg IV over 1 hour every 2 weeks. Treatment continued until there is evidence of disease progression, intolerable toxicity, or other withdrawal criteria are met.
  Participants must be receiving depot octreotide at the time of enrolling into the study. Participants on stable doses of depot octreotide continued to receive the same dose and schedule of their last regimen.
Period: Overall Study
Arm/Group | Carcinoid Tumor | Islet Cell Carcinoma
Started | 31 | 12
Received at Least 1 Dose of Study Drug | 31 | 12
Completed | 25 | 4
Not Completed | 6 | 8
Not completed — Adverse Event | 4 | 4
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Physician Decision | 0 | 2
Not completed — Sponsor Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Carcinoid Tumor: Participants with carcinoid tumor received cixutumumab 10 mg/kg IV over 1 hour every 2 weeks. Treatment continued until there is evidence of disease progression, intolerable toxicity, or other withdrawal criteria are met.
  Participants must be receiving depot octreotide at the time of enrolling into the study. Participants on stable doses of depot octreotide continued to receive the same dose and schedule of their last regimen.
- Islet Cell Carcinoma: Participants received cixutumumab 10 mg/kg IV over 1 hour every 2 weeks. Treatment continued until there is evidence of disease progression, intolerable toxicity, or other withdrawal criteria are met.
  Participants must be receiving depot octreotide at the time of enrolling into the study. Participants on stable doses of depot octreotide continued to receive the same dose and schedule of their last regimen.
- Total: Total of all reporting groups
Arm/Group | Carcinoid Tumor | Islet Cell Carcinoma | Total
Number analyzed (Participants) | 31 | 12 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (9.65) | 61.3 (9.85) | 60.6 (9.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 4 | 21
  Male | 14 | 8 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 29 | 9 | 38
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 30 | 12 | 42
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 31 | 12 | 43

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Progression-Free Survival (PFS) Rate at Six Months
Description: Percentage of participants who are alive and progression-free at 6 month from start of the study treatment over all participants. PFS is defined as the time from the start of study treatment until the date of objectively determined progressive disease (PD) or death due to any cause. Disease progression was assessed via Response Evaluation Criteria in Solid Tumors (RECIST) version 1.0, and defined as at least a 20% increase in the sum of the longest diameters of target lesions, taking as reference the smallest sum longest diameter recorded since the baseline measurements, and/or the appearance of one or more new lesion(s), and/or unequivocal progression of existing nontarget lesions. Participants without documentation of progression or death will be censored at the date of last tumor assessment. The PFS was estimated by the binomial distribution and Kaplan-Meier method.
Time Frame: From Start of Study Treatment to Progressive Disease or Death Due to Any Cause (Up to 6 Months)
Population: All participants who received at least one dose of study drug. Participants censored in the carcinoid tumor arm were 8 and in the islet cell carcinoma arm were 4.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Carcinoid Tumor | Islet Cell Carcinoma
Number analyzed (Participants) | 31 | 12
percentage of participants
  Binomial Distribution; Primary Analysis | 45.2 [27.3 to 64.0] | 41.7 [15.2 to 72.3]
  Kaplan-Meier Method; Secondary Analysis | 54.1 [34.2 to 70.3] | 61.4 [26.6 to 83.5]

2. Secondary Outcome: Percentage of Participants Who Achieve Modified Objective Response Rate (ORR) of Complete Response (CR), Partial Response (PR) and Minor Response (MR) Modified Objective Response Rate (mORR)
Description: Modified ORR is defined as CR+ PR + MR. According to RECIST v1.0, CR was defined as the disappearance of all target and non-target lesions; PR defined as a >30% decrease in the sum of the longest diameters (LD) of the target lesions, taking as reference the baseline sum of the LD and MR defined as 20% - 29% reduction. Disease progression defined as at least a 20% increase in the sum of the longest diameters of target lesions, taking as reference the smallest sum longest diameter recorded since the baseline measurements, and/or the appearance of one or more new lesion(s), and/or unequivocal progression of existing nontarget lesions.
Time Frame: From Start of Treatment Baseline to Disease Progression (Up to 18 Months)
Population: All participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Carcinoid Tumor | Islet Cell Carcinoma
Number analyzed (Participants) | 31 | 12
percentage of participants | 3.2 [0.1 to 16.7] | 0 [0 to 26.5]

3. Secondary Outcome: Percentage of Participants With a Biochemical Response Rate
Description: Determine the biochemical response rate (≥ 50% reduction in tumor-specific markers; may include, not limited to 24 hour urine 5-hydroxyindoleacetic acid, chromogranin A, adrenocorticotropin hormone (ACTH), or gastrin) in the subset of participants with biochemically measurable disease.
Time Frame: From Start of Treatment Up to 18 Months
Population: All participants who received at least one dose of study drug and had evaluable baseline and post-baseline Chromogranin A and Gastrin data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Carcinoid Tumor | Islet Cell Carcinoma
Number analyzed (Participants) | 31 | 12
percentage of participants
  Chromogranin A: number analyzed (Participants) | 25 | 9
  Chromogranin A | 0.0 [0.0 to 13.7] | 22.2 [2.8 to 60]
  Gastrin: number analyzed (Participants) | 6 | 2
  Gastrin | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 84.2]

4. Secondary Outcome: Number of Participants Reporting Treatment-Emergent Adverse Events (TEAEs)
Description: Number of participants that had at least one TEAE is presented. A summary of other non-serious adverse events and all serious adverse events, regardless of causality, is located in the Reported Adverse Events Section.
Time Frame: 18 months
Population: All participants who had received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Carcinoid Tumor | Islet Cell Carcinoma
Number analyzed (Participants) | 31 | 12
Participants | 31 | 12

5. Secondary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) Cycle 1
Time Frame: Prior to the final infusion, immediately after the infusion, and 1, 2, 4, 8, 48, 96, 168, and 336 hours after the completion of the final infusion
Population: Zero participants were analyzed. The assay used to measure serum concentrations of cixutumumab was not fully developed and validated, and the resulting data was therefore not suitable for estimation of PK parameters.
Arm/Group | Carcinoid Tumor | Islet Cell Carcinoma
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: PK: Half-life (t 1/2) Cycle 1
Time Frame: as for outcome 5
Population: as for outcome 5
Arm/Group | Carcinoid Tumor | Islet Cell Carcinoma
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: PK: Area Under Concentration (AUCinf) Cycle 1
Time Frame: as for outcome 5
Population: as for outcome 5
Arm/Group | Carcinoid Tumor | Islet Cell Carcinoma
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: PK: Clearance (CL) Cycle 1
Time Frame: as for outcome 5
Population: as for outcome 5
Arm/Group | Carcinoid Tumor | Islet Cell Carcinoma
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: PK: Volume at Steady State (Vss) Cycle 1
Time Frame: as for outcome 5
Population: as for outcome 5
Arm/Group | Carcinoid Tumor | Islet Cell Carcinoma
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Serum Anti-Cixutumumab Antibody Assessment
Time Frame: 18 months
Population: Zero participants were analyzed due to no data collection due to low number of clinical responses observed.
Arm/Group | Carcinoid Tumor | Islet Cell Carcinoma
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Pharmacodynamics Markers; Concentration of Insulin-like Growth Factor I, II (IGF-I, IGF-II), IGF Body Fat (IGFBF)-1 and IGFBF-2
Time Frame: 18 months
Population: Zero participants were analyzed due to no data collection due to low number of clinical responses observed.
Arm/Group | Carcinoid Tumor | Islet Cell Carcinoma
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Carcinoid Tumor | Islet Cell Carcinoma
Serious Adverse Events (participants affected / at risk) | 12/31 | 6/12
Other Adverse Events (participants affected / at risk) | 31/31 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carcinoid Tumor (N=31) | Islet Cell Carcinoma (N=12)
Deafness (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 0 (0)
Disease progression (General disorders) | 1 (1) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Carcinoid syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Carcinoid Tumor (N=31) | Islet Cell Carcinoma (N=12)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 2 (3)
Deafness (Ear and labyrinth disorders) | 2 (2) | 2 (2)
Ear discomfort (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 2 (2) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Eyelids pruritus (Eye disorders) | 0 (0) | 1 (1)
Metamorphopsia (Eye disorders) | 0 (0) | 1 (1)
Photopsia (Eye disorders) | 5 (5) | 1 (1)
Vision blurred (Eye disorders) | 2 (2) | 1 (1)
Visual impairment (Eye disorders) | 0 (0) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 3 (3) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 9 (20) | 2 (2)
Abdominal pain lower (Gastrointestinal disorders) | 3 (3) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 5 (5) | 3 (3)
Ascites (Gastrointestinal disorders) | 3 (5) | 0 (0)
Constipation (Gastrointestinal disorders) | 5 (7) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 20 (47) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 6 (6) | 2 (2)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 2 (2) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 3 (3) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 1 (1)
Malabsorption (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 14 (23) | 3 (4)
Oral pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 3 (3) | 1 (1)
Vomiting (Gastrointestinal disorders) | 9 (20) | 2 (2)
Asthenia (General disorders) | 5 (8) | 0 (0)
Catheter site erosion (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 3 (4) | 0 (0)
Early satiety (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 20 (36) | 9 (10)
Feeling cold (General disorders) | 0 (0) | 1 (1)
Inflammation (General disorders) | 1 (1) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2) | 1 (1)
Oedema (General disorders) | 2 (2) | 0 (0)
Oedema peripheral (General disorders) | 5 (6) | 2 (2)
Pain (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 4 (5) | 3 (3)
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 (2) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (3) | 0 (0)
Vulval abscess (Infections and infestations) | 1/17 (1) | 0/4 (0)
Contusion (Injury, poisoning and procedural complications) | 6 (8) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (6) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 2 (6) | 3 (3)
Blood alkaline phosphatase increased (Investigations) | 2 (2) | 3 (3)
Blood creatinine increased (Investigations) | 6 (7) | 3 (4)
Blood pressure increased (Investigations) | 0 (0) | 1 (1)
Breath sounds abnormal (Investigations) | 1 (1) | 1 (1)
Clostridium test positive (Investigations) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 3 (3) | 1 (1)
Platelet count decreased (Investigations) | 2 (2) | 0 (0)
Urine output decreased (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 18 (24) | 4 (5)
White blood cell count decreased (Investigations) | 2 (2) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 10 (15) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 6 (7) | 2 (2)
Failure to thrive (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 8 (13) | 6 (11)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (7) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (5) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (12) | 3 (3)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 (6) | 5 (7)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 (5) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 (7) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Disturbance in attention (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 12 (14) | 2 (3)
Dysgeusia (Nervous system disorders) | 4 (5) | 1 (1)
Headache (Nervous system disorders) | 6 (13) | 1 (1)
Tremor (Nervous system disorders) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 4 (5) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (5) | 0 (0)
Nocturia (Renal and urinary disorders) | 2 (2) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary hesitation (Renal and urinary disorders) | 0 (0) | 1 (1)
Penile haematoma (Reproductive system and breast disorders) | 0/14 (0) | 1/8 (1)
Prostatitis (Reproductive system and breast disorders) | 1/14 (1) | 0/8 (0)
Vulvovaginal burning sensation (Reproductive system and breast disorders) | 1/17 (1) | 0/4 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Nail discolouration (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Onychoclasis (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 6 (8) | 2 (3)
Hypertension (Vascular disorders) | 5 (6) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days